CLINICAL TRIAL: NCT04410549
Title: Optical Coherence Tomography for Microvascular Lung Vessels Obstructive Thromboinflammatory Syndrome Assessment in Patients With COVID-19: an Exploratory Study
Brief Title: Pulmonary Optical Coherence Tomography in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Matteo Montorfano, Interventional Cardiology Unit Director, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCT COVID
Record Dates: First submitted 2020-05-21; First posted 2020-06-01 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Pulmonary Embolism
Keywords: COVID-19; PULMONARY EMBOLISM; MICROCLOTS; OCT
MeSH Terms: conditions — COVID-19; Pulmonary Embolism | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 patient with pulmonary thrombosis (Experimental): * patients with COVID-19, high D-dimer levels and contrast CT scan negative for pulmonary thrombosis
  * patients with contrast CT scan positive for pulmonary embolism in areas where contrast CT scan was negative.
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT)

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography (OCT) — To perform OCT in pulmonary artery of patient with COVID-19

SUMMARY:
To evaluate by intravascular OCT study the presence of microvascular pulmonary thrombosis in patients with COVID-19, high D-dimer levels and contrast CT scan negative for pulmonary thrombosis. We'll also evaluate the extension of microvascular pulmonary thrombosis in patients with contrast CT scan positive for pulmonary embolism in areas where contrast CT scan was negative.

DETAILED DESCRIPTION:
Background:Severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2) infection represents a pandemic emergency of dramatic proportions. The clinical course of SARS-CoV-2 infection often meets the criteria for acute respiratory distress syndrome (ARDS), with progressive severity ultimately leading to a rapid death. It appeared that the progressive worsening lung function of patients infected with SARS-CoV-2 was potentially driven by host immune response. SARS-CoV-2 replication in lung epithelial cells causes direct cellular damage and release of pro-inflammatory alarmins from dying cells. The successive complement system activation causes massive local release of pro-inflammatory cytokines and consequent severe collateral tissue injury and massive vascular endothelial and alveolar epithelial cell damage and microvascular thrombosis. Functional implications of this peculiar ARDS pathogenesis include a progressive worsening of ventilation/perfusion imbalances and a loss of hypoxic vasoconstriction reflexes, with a marked component of microvascular pulmonary thrombosis, as suggested by lactate dehydrogenase and D-dimer elevations. In the late stages of ARDS, the progression of endothelial damage with microvascular thrombosis can spread locally in the lung and potentially extends the systemic inflammatory reaction involving the microvascular bed of the kidneys, brain and other vital organs. A new mechanism of lung damage was recently proposed, with dramatic alveolar endothelial damage leading to a progressive endothelial pulmonary syndrome with microvascular thrombosis and suggests MicroCLOTS (microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome) as an atypical ARDS working hypothesis. In fact, thromboembolic events rate in COVID-19 patients appears not negligible, and a prophylactic utilization of low molecular weight heparin (LMWH) should be considered.Several biomarkers are under investigation to better determine the risk of thromboembolic events and to determine the patients who could benefit more of a prophylactic therapy with LMWH. Among others, D-Dimer is often elevated in COVID-19 patients and should be used as the most important parameter for thromboembolic risk stratification, together with other inflammation index like C-reactive-protein, interleukin 6 (IL-6) and ferritin. Nevertheless, a not negligible part of patient with COVID-19 pneumonia presents high D-dimer level with computed tomography (CT) scan negative for pulmonary embolism. Despite these patients could presents pulmonary microvascular thrombosis (MicroCLOTS), it has never been proven and an aggressive anticoagulant treatment is currently not utilized. A diagnostic technique more sensible than the CT scan on the small pulmonary arteries could theoretically allow the detection of MicroCLOTS thus justifying a more aggressive anticoagulant regimen.

Optical coherence tomography:The optical coherence tomography (OCT) is a near-infrared light source-based imaging technique with a resolution of 10-20 um. It acquires longitudinal sequences of cross-sectional images (100 frames/s) in a blood-free environment, resulting in sharp border definition between lumen and vessel wall. It is routinely used in percutaneous coronary intervention (PCI) to better characterize vessel anatomy, as well as ascertainment of full stent deployment and expansion. Moreover, OCT has been shown to have a good correlation with histology even in the evaluation of pulmonary artery morphology, particularly in the evaluation of pulmonary arterial wall thickness. Furthermore, OCT has been used to better characterized distal Type Chronic Thromboembolic Pulmonary Hypertension, and to guide its treatment with percutaneous transluminal pulmonary angioplasty. Hong et al evaluated with OCT three patients who were highly suspected for peripheral pulmonary arteries thrombi but had negative CT scan for pulmonary embolism. Thrombi were found in most of imaged vessels in these patients. Red and white thrombi can be differentiated, according to features of the thrombus on OCT images. After anticoagulation treatment, these patients' symptoms and hypoxemia improved. Repeated OCT imaging showed that most thrombi disappeared or became smaller. OCT was also used in evaluation of pulmonary arterial vasculopathy in Systemic Sclerosis, showing an unexpected evidence of pulmonary artery thrombus formation in 19% of systemic-sclerosis patients with pulmonary arterial hypertension.

There are sufficient data showing OCT to be a useful tool to identify intravascular thrombi in patients with chronic thromboembolic pulmonary hypertension, together with an increase in vessel wall thickness in most patients with pulmonary hypertension.

Aim of the study:To evaluate by intravascular OCT study the presence of microvascular pulmonary thrombosis in patients with COVID-19, high D-dimer levels and contrast CT scan negative for pulmonary thrombosis. Investigators will also evaluate the extension of microvascular pulmonary thrombosis in patients with contrast CT scan positive for pulmonary embolism in areas where contrast CT scan was negative.

Inclusion Criteria (part A): 1) Severe pulmonary coronarvirus disease 19 (COVID 19) with suspect for MicroCLOTS (microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome) AND 2) Contrast CT scan negative for pulmonary thrombosis AND 3) D-Dimer > 10 mcg/mL OR 4) 5 < D-dimer < 10 mcg/mL and either C Reactive Protein (CRP) > 100 mg/dL or IL-6 > 6 pg/mL or ferritin > 900 ng/L; (part B): 1) Severe pulmonary coronarvirus disease 19 (COVID 19) with suspect for MicroCLOTS (microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome) AND 2) Contrast CT scan positive for pulmonary thrombosis

Exclusion Criteria: 1) Age < 18 2) Pregnancy or breastfeeding 3) Known allergy to iodinated contrast dye 4) Hemodynamic instability 5) Glomerular Filtration rate < 30 ml/min 6) Active bleeding or absolute contraindication to anticoagulant therapy

OCT procedure: Femoral vein echo-guided puncture; 6 Fr 11 cm sheath insertion; Unfractionated heparin administration (70 - 100 U/kg) to achieve an activated clotting time (ACT) between 250 and 300 seconds; Pulmonary artery cannulation with 5 Fr Multipurpose (MP) catheter (Cordis, Dublin, Ohio) and Storq wire (Cordis); Pulmonary artery pressure measurement; Selective pulmonary artery cannulation and angiography (The choice of the pulmonary arteries to be cannulated will be driven by "ground glass" area at CT scan); 5Fr MP catheter will be changed for 6Fr MP guiding catheter over the Storq wire; Storq wire removal and 0.014" Balance wire distally advanced; OCT images acquisition (In order to remove all the blood, as well as to obtain clear images, iodinated contrast is infused at a flow rate of 5 mL/s over 4 s, at 400 psi of pressure (Acist, Eden Prairie, Minnesota). Automatic pullback at 20 mm/s); If needed, blood samples can be taken through Recover catheter (Hexacath, Rueil-Malmaison, France).

The same procedure will be performed: on "healthy" (without ground glass appearance at CT scan) area in the same lung and on contralateral lung, both in "ground glass" and "healthy" areas according to CT scan.

PRIMARY ENDPOINT: 1) Overall safety of OCT procedure in COVID-19 pneumonia patients 2) Presence of microvascular pulmonary thrombosis at OCT assessment in COVID-19 patients, both in "ground glass" and "healthy" ventilated areas.

SECONDARY ENDPOINT: 1) Pulmonary artery vessel anatomy characterization in COVID-19 patients 2) Correlations with single trans-thoracic echocardiography (TTE) pulmonary hypertension (PH, estimated systolic pulmonary artery pressure > 35 mmHg) and right ventricular disfunction (RVD: tricuspid annular plane systolic excursion < 17 mm or Doppler tissue imaging S wave < 9.5 cm/sec) 3) Dynamic correlations with standard inflammatory, coagulation and tissue damage biomarkers: CRP, ferritin, D-dimer, NT-proBNPO, troponins, LDH)

Study design, sample size, statistical analysis: The study is an open label, prospective, interventional clinical study of the safety, tolerability and potential diagnostic value of optical coherence tomography for microvascular lung vessels obstructive thromboinflammatory syndrome assessment in patients with COVID-19 pneumonia.

This is an exploratory study and will be conducted in 10 patients with mild-to-severe ARDS. The sample size calculation was designed for safety assessment based on a reference population of last 100 patients who underwent OCT at our Institution for coronary Artery Disease (CAD) in which a rate of SAEs lower than 1% have been recorded (personal communication)

Primary endpoint: As for safety analysis, the number of ADR (expected/unexpected) and SAEs (expected/unexpected and/or related/not related) and the percentage of subjects experiencing ADR and SAEs in the study will be summarized by severity and within body system involved. Narratives will also be presented.

Secondary endpoints: Continuous variables will be summarized with indices of location (i.e. mean or median) and dispersion (i.e. standard deviation or interquartile range), as appropriate. All relevant estimates will be reported with the corresponding 95% Confidence Intervals (CI).

The time to event endpoints will be described using the Kaplan-Meier approach and estimates at pre-defined time points will be obtained along with 95%Cis. Patients will be censored at study closure, withdrawn of consent or loss to follow-up.

Subgroup analyses and regression models (i.e. logistic model on proportions and Cox model on time to event outcomes) will be performed considering age, sex, biological features.

Withdrawal and Premature Termination or Suspension of Study Investigators may terminate a study subject's participation in the study if: any clinical AE, or other medical condition or situation occurs such that continued participation in the study would not be in the best interest of the subject, the subject meets an exclusion criterion, either newly developed or not previously recognized (except those caused by ARDS and SARS-CoV-2 infection), that precludes further study participation; this study may be suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided.

Fundings: not appropriate. The procedure will be charged to SSN as a diagnostic procedure applied to patients clinically suspected of microCLOTS in COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

(part A)

* Severe pulmonary coronarvirus disease 19 (COVID 19) with suspect for MicroCLOTS (microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome) AND
* Contrast CT scan negative for pulmonary thrombosis AND
* D-Dimer > 10 mcg/mL OR
* 5 < D-dimer < 10 mcg/mL and either C Reactive Protein (CRP) > 100 mg/dL or IL-6 > 6 pg/mL or ferritin > 900 ng/L

(part B)

* Severe pulmonary coronarvirus disease 19 (COVID 19) with suspect for MicroCLOTS (microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome) AND
* Contrast CT scan positive for pulmonary thrombosis

Exclusion Criteria:

* Age < 18
* Pregnancy or breastfeeding
* Known allergy to iodinated contrast dye
* Hemodynamic instability
* Glomerular Filtration rate < 30 ml/min
* Active bleeding or absolute contraindication to anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
optical coherence tomography pulmonary microthrombosis assessment in COVID-19 pneumonia patients | through study completion, an average of 1 month
  Study primary endpoints will be evaluation of OCT procedure overall safety in COVID-19 pneumonia patients and assessment of the presence of microvascular pulmonary thrombosis in COVID-19 patients, both in "ground glass" and "healthy" ventilated areas.

SECONDARY OUTCOMES:
Pulmonary artery vessel anatomy characterization | through study completion, an average of 1 month
  Pulmonary artery vessel anatomy characterization in COVID-19 pneumonia patients through OCT diagnostic technique
  * Correlations with single trans-thoracic echocardiography (TTE) pulmonary hypertension (PH, estimated systolic pulmonary artery pressure > 35 mmHg) and right ventricular disfunction (RVD: tricuspid annular plane systolic excursion < 17 mm or Doppler tissue imaging S wave < 9.5 cm/sec).
  * Dynamic correlations with standard inflammatory, coagulation and tissue damage biomarkers: CRP, ferritin, D-dimer, NT-proBNPO, troponins, LDH)
Correlation between TTE pulmonary hypertension and right ventricular disfunction | through study completion, an average of 1 month
  Correlations with single trans-thoracic echocardiography (TTE) pulmonary hypertension (PH, estimated systolic pulmonary artery pressure > 35 mmHg) and right ventricular disfunction (RVD: tricuspid annular plane systolic excursion < 17 mm or Doppler tissue imaging S wave < 9.5 cm/sec)
Correlations with standard inflammatory, coagulation and tissue damage | through study completion, an average of 1 month
  Pneumonia COVID-19 dynamic correlation with inflammation and coagulation markers

CONTACTS AND LOCATIONS:
Locations (2):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciceri F, Beretta L, Scandroglio AM, Colombo S, Landoni G, Ruggeri A, Peccatori J, D'Angelo A, De Cobelli F, Rovere-Querini P, Tresoldi M, Dagna L, Zangrillo A. Microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome (MicroCLOTS): an atypical acute respiratory distress syndrome working hypothesis. Crit Care Resusc. 2020 Apr 15;22(2):95-97. doi: 10.51893/2020.2.pov2. Online ahead of print. PMID 32294809
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299
- [Background] Wijns W, Shite J, Jones MR, Lee SW, Price MJ, Fabbiocchi F, Barbato E, Akasaka T, Bezerra H, Holmes D. Optical coherence tomography imaging during percutaneous coronary intervention impacts physician decision-making: ILUMIEN I study. Eur Heart J. 2015 Dec 14;36(47):3346-55. doi: 10.1093/eurheartj/ehv367. Epub 2015 Aug 4. PMID 26242713
- [Background] Li N, Zhang S, Hou J, Jang IK, Yu B. Assessment of pulmonary artery morphology by optical coherence tomography. Heart Lung Circ. 2012 Dec;21(12):778-81. doi: 10.1016/j.hlc.2012.07.014. Epub 2012 Aug 10. PMID 22884790
- [Background] Hong C, Wang W, Zhong NS, Zeng GQ, Wu H. Using optical coherence tomography to detect peripheral pulmonary thrombi. Chin Med J (Engl). 2012 Sep;125(17):3171-4. PMID 22932201
- [Background] Schwaiger JP, Loder CD, Dobarro D, Kaier T, Reddecliffe S, Schreiber BE, Handler C, Denton CP, Coghlan JG. Optical coherence tomography evaluation of pulmonary arterial vasculopathy in Systemic Sclerosis. Sci Rep. 2017 Feb 24;7:43304. doi: 10.1038/srep43304. PMID 28233825
- [Background] Dai Z, Fukumoto Y, Tatebe S, Sugimura K, Miura Y, Nochioka K, Aoki T, Miyamichi-Yamamoto S, Yaoita N, Satoh K, Shimokawa H. OCT imaging for the management of pulmonary hypertension. JACC Cardiovasc Imaging. 2014 Aug;7(8):843-5. doi: 10.1016/j.jcmg.2014.01.020. No abstract available. PMID 25124017
- [Background] van der Sijde JN, Karanasos A, van Ditzhuijzen NS, Okamura T, van Geuns RJ, Valgimigli M, Ligthart JM, Witberg KT, Wemelsfelder S, Fam JM, Zhang B, Diletti R, de Jaegere PP, van Mieghem NM, van Soest G, Zijlstra F, van Domburg RT, Regar E. Safety of optical coherence tomography in daily practice: a comparison with intravascular ultrasound. Eur Heart J Cardiovasc Imaging. 2017 Apr 1;18(4):467-474. doi: 10.1093/ehjci/jew037. PMID 26992420
- [Derived] Hajjar LA, Ancona MB, Filho RK, Tresoldi M, Caldas JG, Monti G, Carnevale FC, De Cobelli F, Moreira de Assis A, Ciceri F, Landoni G, Dijkstra J, Moroni F, Abizaid AAC, Willemann Ungaretti F, Carvalho Carmona MJ, De Backer D, Pompilio CE, de Britto FS Jr, Campos CM, Zangrillo A, Montorfano M. Microvascular lung vessels obstructive thromboinflammatory syndrome in patients with COVID-19: Insights from lung intravascular optical coherence tomography. Front Med (Lausanne). 2023 Feb 16;10:1050531. doi: 10.3389/fmed.2023.1050531. eCollection 2023. PMID 36873865

DOCUMENTS (1):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT04410549/Prot_000.pdf